CLINICAL TRIAL: NCT04128462
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase 3 Study to Evaluate the Efficacy, Safety, and Tolerability of MNK6105 (an Intravenous Formulation of L-Ornithine Phenylacetate) in Hospitalized Patients With Cirrhosis and Hyperammonemia Associated With an Episode of Hepatic Encephalopathy
Brief Title: MNK-6105 for Patients With Cirrhosis and High Ammonia Levels Affecting Brain Function
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Business Decision
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MNK61053106; 2019-001635-31 (EudraCT Number)
Record Dates: First submitted 2019-10-14; First posted 2019-10-16 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Hepatic Encephalopathy
Keywords: Overt HE diagnosis
MeSH Terms: conditions — Hepatic Encephalopathy | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MNK6105 + SoC (Experimental): Participants will receive standard of care (SoC), along with MNK-6105 delivered by continuous intravenous (IV) infusion as follows:
  * Loading dose: 20 g infused over 6 hours
  * Intermediate dose: 15 g infused over 18 hours
  * Maintenance dose: 15 g infused over 24 hours for up to 4 days
  Interventions: Drug: MNK-6105; Drug: Standard of Care
- Placebo + SoC (Placebo Comparator): Participants will receive SoC, along with continuous IV infusion of matching placebo for 5 days.
  Interventions: Drug: Placebo; Drug: Standard of Care

INTERVENTIONS:
Drug: MNK-6105 — L-Ornithine Phenylacetate for IV infusion
  Other Names: L-Ornithine Phenylacetate
  Arms: MNK6105 + SoC
Drug: Placebo — Matching placebo for IV infusion
  Other Names: Matching Placebo
  Arms: Placebo + SoC
Drug: Standard of Care — Lactulose ± rifaximin as SoC treatment for overt HE should be administered per the clinical judgement of the investigator and usual institutional practice.
  Other Names: SoC

SUMMARY:
This study is for patients with cirrhosis and hepatic encephalopathy who are in the hospital. This means they have a high ammonia level which is affecting their brain function.

All patients will receive the standard of (regular) care. Each will have an equal chance (like flipping a coin) of receiving the experimental drug or placebo along with the standard care.

Each patient will have tests during the first 24 hours, receive treatment for up to 5 days, and have 30 days of follow-up.

ELIGIBILITY:
Inclusion Criteria:

To be included, a patient must:

* Be the age of majority in their country (considered an adult)
* Be male or non-pregnant, non-lactating female
* Have OHE (Stage 2, 3, or 4) as a complication of cirrhosis
* Have been hospitalized within 24 hours before start of infusion (SOI)
* Receive at least 6 hours of SoC treatment

Exclusion Criteria:

Patients will be excluded if they have inadequate renal function or any other disease, laboratory value, or condition (including allergy, drug use or treatments) that per protocol or in the opinion of the investigator, might increase the risk of compromising:

1. health or well-being of the patient
2. safety of study staff
3. analysis of results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Number of patients with a clinical response at Day 5 | at Day 5 (within 36 months)

SECONDARY OUTCOMES:
Number of patients discharged 30 days after end of treatment. | at Day 35 (within 36 months)
Number of patients readmitted to the hospital due to overt hepatic encephalopathy (OHE) 30 days after discharge. | 30 days after discharge (within 36 months)
Number of patients with adverse events or deaths during the study | within 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Team Leader, Study Director — Mallinckrodt

IPD SHARING:
Plan to Share IPD: No